CLINICAL TRIAL: NCT01037179
Title: An Open-Label, Long-Term Study With AL-4943A Ophthalmic Solution, 0.2% in Patients With Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-09-050
Record Dates: First submitted 2009-12-18; First posted 2009-12-22 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL-4943A (Experimental): Olopatadine Hydrochloride Ophthalmic Solution, 0.2%, 2 drops instilled in each eye twice daily for 10 weeks
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%
  Other Names: PATADAY®

SUMMARY:
The objective of this study is to assess safety and efficacy of long-term use of AL-4943A (Olopatadine Hydrochloride Ophthalmic Solution, 0.2%) in patients with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written consent.
* Subjects must have a diagnosis of allergic conjunctivitis.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Itching and/or hyperemia associated with diseases other than allergic conjunctivitis.
* Retinal detachment, diabetic retinopathy, or any progressive disease in posterior segment of the eye.
* Known history of ocular infection.
* Contact lens wear during study.
* Pregnant, nursing.
* Participation in another clinical study within 30 days of Informed Consent.
* Other protocol-defined exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Mean Itching Score by Visit | Up to Week 10
  Ocular itching will be assessed by the subject and graded on a 6-point scale, where 0=did not occur and 5=virtually all the time over the past 3 days.
Mean Total Hyperemia Score by Visit | Up to Week 10
  Ocular hyperemia (redness) will be assessed by the investigator. Total hyperemia score is defined as the sum of the palpebral and bulbar conjunctival scores.

SECONDARY OUTCOMES:
Mean Subjective Symptoms by Visit | Up to Week 10

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Center, Osaka, Osaka, Japan